CLINICAL TRIAL: NCT02526654
Title: Validation and Reproducibility of the Heidelberg Edge Perimeter in the Detection of Visual Field Defects in Glaucomatous Patients
Brief Title: Heidelberg Edge Perimetry (HEP) Detecting Glaucomatous Visual Field Defects
Acronym: HEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-340
Record Dates: First submitted 2015-07-30; First posted 2015-08-18 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glaucoma Subjects (Experimental): Subjects with glaucoma were recruited based on characteristic glaucomatous disc damage and visual field changes. They will perform visual field with Heidelberg Edge Perimeter and Octopus visual field. Optical Coherence Tomography will image the retinal nerve fiber layer.
  Interventions: Diagnostic Test: Heidelberg Edge Perimeter; Diagnostic Test: Octopus Visual Field; Diagnostic Test: Optical Coherence Tomography
- Healthy Controls (Experimental): Subjects that do not have glaucoma and are recruited for testing will perform visual field with Heidelberg Edge Perimeter and Octopus visual field. Optical Coherence Tomography will image the retinal nerve fiber layer.
  Interventions: Diagnostic Test: Heidelberg Edge Perimeter; Diagnostic Test: Octopus Visual Field; Diagnostic Test: Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: Heidelberg Edge Perimeter — HEP measures peripheral vision
  Other Names: HEP
Diagnostic Test: Octopus Visual Field — OVF measures peripheral vision
  Other Names: OVF
Diagnostic Test: Optical Coherence Tomography — OCT measures retinal nerve fiber layer thickness
  Other Names: OCT

SUMMARY:
The purpose of this study is to compare standard automated perimetry (SAP) using the Heidelberg Edge Perimeter (HEP) to the Octopus Visual Field (OVF) analyzer and determine test-retest reliability of both parameters in detecting glaucomatous visual field losses. This study will also investigate novel imaging parameters of the optic nerve head and new automated structure-function reports.

DETAILED DESCRIPTION:
Each participant undergo the following tests:

1. Standard ophthalmic examination (usual care): Best-corrected visual acuity, biomicroscopy (look at front of eye), intraocular pressure (IOP) using Goldman applanation tonometry, central corneal thickness measurement and fundoscopy (look at back of eye).
2. Octopus Visual Field (OVF) Analyzer using G-top strategy recording mean deviation (MD) and pattern standard deviation (PSD).
3. Heidelberg Edge Perimeter (HEP) standard automated perimetry (SAP) using advanced staircase thresholding algorithm (ASTA).
4. Spectralis optical coherence tomography (OCT) using glaucoma module premium edition (GMPE) software to measure minimum rim width (MRW) and retinal nerve fiber layer (RNFL) thickness in 6 sectors (superior nasal, superior temporal, inferior nasal, inferior temporal, nasal and temporal) in the retina.

Order of HEP SAP III and OVF, and order of the eye tested (right vs. left) if both eyes of patients meet inclusion criteria will be randomized. Patients with glaucoma will be randomly chosen and asked to return in 3 to 6 months for repeat HEP and OVF testing.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Best corrected visual acuity of 20/40 or better in the tested eye.
* Spherical refraction within ±5.0 D, and cylinder correction within ±3.0 D.
* History of glaucoma, defined as:
* Characteristic of glaucomatous disc damage: (local narrowing, notching, or absence of the neuroretinal rim in the absence of disc pallor elsewhere).

Exclusion Criteria:

* Any condition preventing adequate examination of the pupil or visual field testing (e.g. ptosis, dense corneal opacities or lens opacities);
* Active infection of the anterior or posterior segments of the eye;
* Any intraocular surgical or laser procedure within the previous 4 weeks;
* Participants taking a medication known to affect visual field sensitivity, a coexisting intraocular disease affecting visual field, or a problem other than glaucoma affecting color vision will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Katz, MD, Principal Investigator — Wills Eye Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cui QN, Fudemberg SJ, Resende AF, Vu TA, Zhou C, Rahmatnejad K, Hark LA, Myers JS, Katz LJ, Waisbourd M. Validation of the structure-function correlation report from the heidelberg edge perimeter and spectral-domain optical coherence tomography. Int Ophthalmol. 2019 Mar;39(3):533-540. doi: 10.1007/s10792-018-0836-z. Epub 2018 Feb 2. PMID 29396688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Glaucoma Service at Wills Eye Hospital between December 2014 and June 2015. Healthy controls were recruited from staff, family and friends.
Pre-assignment Details: Before study tasks, Informed Consent was conducted and obtained according to the International Conference on Harmonization Good Clinical Practices (ICH GCP) guidelines with opportunity for all questions to be answered.
Groups:
- Glaucoma Subjects: Subjects with glaucoma were recruited based on characteristic glaucomatous disc damage and visual field changes.
- Healthy Controls: Healthy subjects that do not have glaucoma and have no other eye diseases.
Period: Overall Study
Arm/Group | Glaucoma Subjects | Healthy Controls
Started | 79 | 36
Completed | 79 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Glaucoma Subjects: Subjects with glaucoma were recruited based on characteristic glaucomatous disc damage and visual field changes from the Glaucoma Service at Wills Eye Hospital in Philadelphia, Pennsylvania. They will perform visual field with Heidelberg Edge Perimeter and Octopus visual field. Optical Coherence Tomography will image the retinal nerve fiber layer.
- Healthy Controls: Healthy control subjects that do not have glaucoma and are recruited for testing will perform visual field with Heidelberg Edge Perimeter and Octopus visual field from staff, family and friends of the Glaucoma Service at Wills Eye Hospital in Philadelphia, Pennsylvania. Optical Coherence Tomography will image the retinal nerve fiber layer.
- Total: Total of all reporting groups
Arm/Group | Glaucoma Subjects | Healthy Controls | Total
Number analyzed (Participants) | 79 | 36 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 47
  >=65 years | 56 | 12 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 23 | 69
  Male | 33 | 13 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 15 | 36
  White | 55 | 17 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 79 | 36 | 115

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient Between HEP and OVF Mean Deviation (MD)
Description: Pearson's correlation coefficient between Heidelberg Edge Perimeter (HEP) and Octopus Visual Field (OVF) Mean Deviation (MD) for glaucoma patients and controls to determine if HEP can detect glaucoma as well as OVF. The closer the values of both parameters for both machines, the better comparable the two machines are to each other in detecting glaucoma.
Time Frame: Baseline visit, 1 hour
Measure: Number; unit: Pearson's correlation coefficient
Groups:
- Glaucoma Subjects: 79 glaucoma subjects defined by characteristic glaucomatous disc damage and visual field changes
- Healthy Controls: 36 healthy control subjects with no glaucoma or other eye diseases.
Arm/Group | Glaucoma Subjects | Healthy Controls
Number analyzed (Participants) | 79 | 36
Pearson's correlation coefficient | -.86 | -.37

2. Secondary Outcome: Repeatability of Optical Coherence Tomography (OCT) Parameters
Description: A subgroup of participants were randomly selected to return at 3 and 6 months for repeat testing. Not all eyes were included. Repeatability of optical coherence tomography (OCT) to consistently detect minimum rim width (MRW) global thickness will be assessed by Pearson's interclass correlation coefficients (ICC). A larger ICC indicates measurements have greater repeatability. Greater than 0.75 indicated excellent repeatability; 0.40 to 0.75 indicated fair to good, and less than 0.40 indicated poor reliability.
Time Frame: Month 6 visit, 1 hour
Population: not all eyes were included in this sub- analysis. inconclusive results were not included.
Measure: Number (95% Confidence Interval); unit: Intraclass correlation coefficients
Units Other Than Participants: eyes
Groups:
- Glaucoma Subjects: 36 eyes from 30 glaucoma patients were analyzed.
- Healthy Controls: 59 eyes from 30 healthy controls were analyzed.
Arm/Group | Glaucoma Subjects | Healthy Controls
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 36 | 59
Intraclass correlation coefficients | .99 [.99 to 1.00] | .99 [0.99 to 1.00]

3. Secondary Outcome: Correlations Between Structure-function Automated Report and Clinical Impression
Description: Heidelberg Edge Perimeter (HEP) Visual Field (VF) and spectral domain optical coherence tomography (SD OCT) printouts from only the glaucoma subgroup were assessed. Retinal Nerve Fiber Layer (RNFL) and Minimum Rim Width (MRW) from SD OCT and HEP VF automated reports were compared to the clinical interpretations by 3 glaucoma specialists.
Time Frame: Baseline visit, 1 hour
Population: Not all eyes (automated reports) met inclusion criteria. Healthy control eye were was not included in this portion of the study. Only glaucoma subgroup received clinical interpretations by 3 glaucoma specialists.
Measure: Number (95% Confidence Interval); unit: Kappa
Units Other Than Participants: eyes
Groups:
- Glaucoma Subjects: 53 eyes from 45 subjects with glaucoma characterized by glaucomatous disc and visual field damage.
Arm/Group | Glaucoma Subjects
Number analyzed (Participants) | 45
Number analyzed (eyes) | 53
Kappa | 0.62 [.54 to .70]

ADVERSE EVENTS:
Time Frame: eye examination, 1 hour
Groups:
- Healthy Controls: Healthy control subjects that do not have glaucoma or other eye diseases.
Arm/Group | Glaucoma Subjects | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/36
Other Adverse Events (participants affected / at risk) | 0/79 | 0/36

LIMITATIONS AND CAVEATS:
Small sample size and varied severity of disease in the glaucoma group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No